CLINICAL TRIAL: NCT03696134
Title: Investigating Musculoskeletal Health and Wellbeing: A Cohort Study
Brief Title: Investigating Musculoskeletal Health and Wellbeing
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 17113
Record Dates: First submitted 2018-09-17; First posted 2018-10-04 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Musculoskeletal Pain, Frailty, Disability
MeSH Terms: conditions — Musculoskeletal Pain; Frailty | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnaire

SUMMARY:
Background The progression and associations of central and peripheral musculoskeletal pain, frailty, disability and fracture risks are not well known. This study aims to characterise the development and progression of different frailty, pain and disability phenotypes and their individual associations.

Methods A prospective cohort of 10000 people aged > 18 will be recruited from general practice surgeries, secondary care and the general public. Data collection waves will be at baseline,and then annual follow-ups for up to five years. Data will be collected using a questionnaire asking about demographic characteristics, pain severity (0-10 scales), pain distribution (a pain Mannikin), pain quality (the McGill Pain Questionnaire), central pain (the CAP-Knee Scale), fracture risks (a modified version of the FRAX instrument), frailty (the Fried Criteria and the FRAIL scale) and disability (the FRAIL scale).

Discussion Participant data will be analysed to determine phenotypic subgroups of frailty, pain and disability. Further to this, the progression of these characteristics and their influences upon health and wellbeing will be quantified.

ELIGIBILITY:
Inclusion Criteria:

- Ability to give informed consent. Aged 18 and over Frailty score of ≥ 0.12 on the eFI Have or are at risk of developing musculoskeletal frailty, pain or disability

Exclusion Criteria:

- Inadequate understanding of verbal explanations or written information in English; Special communication needs; Receiving dialysis; Receiving home oxygen; Terminal cancer; Unstable angina or heart failure; Serious mental illness; Dementia.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a broad range of sources, including the community, primary and secondary care health services. Diverse recruitment pathways will enable enrichment of the cohort with participants from a range of backgrounds and suitable for a range of potential interventions aiming to reduce frailty, pain or disability. Participants may be recruited from GP surgeries, community based clinics, Musculoskeletal Pathway (Physiotherapy and occupational health clinics in primary care), hospital patient waiting lists, hospital outpatients' lists and physiotherapy services, or as participants from previous studies undertaken by the University of Nottingham or Nottingham University Hospitals NHS Trust who have expressed an interest in future research, and people who respond to online material.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-06-22 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Presence, severity and prevalence of frailty, as measured by response to the study questionnaire at annual intervals | 5 years
  Frailty will be classified using the 5-item FRAIL scale (Fatigue, Resistance, Ambulation, Illnesses, & Loss of Weight).
Presence and prevalence of pain | 5 years
  Pain distribution will be recorded in a pain manikin.
Presence and prevalence of disability | 5 years
  Disability will be determined using the five Fried Criteria modified for questionnaire delivery.

SECONDARY OUTCOMES:
1. Classification of phenotypic subgroups | 5 years
  Demographic characteristics will be recorded; age at baseline, sex, race, socioeconomic position (deprivation index, urban/rural indicators will be derived from postcode data), smoking habits, weight, height and alcohol consumption. Fracture risk will be assessed using a modified version of the FRAX instrument (substituting secondary osteoporosis for self-reported osteoporosis and without using data for bone mineral density measurements).
2. Classification of comorbid conditions | 5 years
  Co-morbidities will be assessed using the Charlson Comorbidity Index
3. Medication usage | 5 years
  Participants will self-report their current medications (prescribed and over the counter).
4. Identification of potential research participants | 5 years
  The Charlson Comorbidity Index
Prevalence of Comorbid conditions | 5 years
  the count of comorbidities
Classification of Rheumatic Comorbid conditions | 5 years
  Rheumatic Disease Comorbidity Index (RDCI).

CONTACTS AND LOCATIONS:
Overall Officials: David Walsh, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Background] Millar B, McWilliams DF, Abhishek A, Akin-Akinyosoye K, Auer DP, Chapman V, Doherty M, Ferguson E, Gladman JRF, Greenhaff P, Stocks J, Valdes AM, Walsh DA. Investigating musculoskeletal health and wellbeing; a cohort study protocol. BMC Musculoskelet Disord. 2020 Mar 21;21(1):182. doi: 10.1186/s12891-020-03195-4. PMID 32199451
- [Derived] Chaplin WJ, McWilliams DF, Millar BS, Gladman JRF, Walsh DA. The bidirectional relationship between chronic joint pain and frailty: data from the Investigating Musculoskeletal Health and Wellbeing cohort. BMC Geriatr. 2023 May 5;23(1):273. doi: 10.1186/s12877-023-03949-4. PMID 37147635